CLINICAL TRIAL: NCT04230980
Title: The Use of Gabapentin for Post-Operative Pain Control and Narcotic Reduction in Scrotal Surgery
Brief Title: Gabapentin for Post-Operative Pain Control and Narcotic Reduction in Scrotal Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-08020686
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Results first posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Non-obstructive Azoospermia
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Gabapentin (Experimental): Participants receive Gabapentin 600mg tablet taken pre-operatively and 300mg taken three times a day for 3 days.
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): Participants receive Placebo tablet taken pre-operatively and three times a day for 3 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — Gabapentin 600mg tablet
  Arms: Gabapentin
Drug: Placebo — Placebo tablet
  Arms: Placebo

SUMMARY:
The use of non-narcotic multi-modal analgesia to be used in the pre-operative, peri-operative and post-operative period to reduce or potentially eliminate narcotic usage following scrotal surgery. Research study results have shown that the use of anti-inflammatories in the peri-operative period reduces both pain and narcotic use. The hypothesis is that adding another agent in the multi-modal pathway will further reduce pain and potentially reduce narcotic usage.

DETAILED DESCRIPTION:
This is a double-blinded, placebo-controlled, randomized trial that will recruit patients categorized into two study arms. Patients in the gabapentin arm will receive gabapentin 600mg taken pre-operatively and 300mg taken three times a day for 3 days, while patients in the placebo arm will receive a placebo drug taken pre-operatively three times a day for 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants undergoing microsurgical testicular sperm extraction.
* Participants over 18 years of age who can provide informed consent
* Participants with no contraindication to the consumption gabapentin or documented allergy/intolerance
* Participants not currently using opiates for another reason

Exclusion Criteria:

* Contraindication to the consumption of celecoxib or gabapentin
* History of substance abuse (including prior opiate abuse)
* Narcotic use within last 3 months
* Any of the following comorbidities: renal failure, heart disease, peptic ulcer disease, cerebrovascular disease, significant liver disease, untreated depression, chronic pain disorder, or bleeding diatheses
* Medical history or concurrent illness that the investigator considers sufficiently serious to interfere with the conduct, completion, or results of this trial, or constitutes an unacceptable risk to the subject

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Gal, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gabapentin | Placebo
Started | 36 | 38
Completed | 35 | 35
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: 1 subject on the gabapentin arm and 3 subjects on the placebo arm were excluded as data collected from these participants was insufficient for analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Placebo | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (10.1) | 34.9 (7.1) | 36.5 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 35 | 35 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 25 | 26 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Pain Score as Measured by the NRS-11 Scale
Description: The Numerical pain Rating Scale (NRS-11) is an 11-point numerical pain rating scale used to measure levels of pain. The lowest possible score is 0 with 0 meaning no pain, and the highest possible score is 10 with 10 meaning severe pain.
Time Frame: Post-operative day 0 (the day of surgery, after surgery was completed) through post-operative day 7
Population: 1 subject has been lost to followup in the gabapentin arm and was therefore excluded from analysis. 2 subjects have been lost to followup in the placebo arm and were therefore excluded from analysis. 1 subject experienced an adverse event in the placebo arm and was taken off the study medication and was therefore excluded from analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 35 | 35
scores on a scale
  Post-Operative Day 0 | 1.91 (1.63) | 3.05 (2.68)
  Post-Operative Day 1, midnight | 2.27 (1.55) | 3.24 (2.7)
  Post-Operative Day 1, before noon | 2.02 (1.8) | 3.33 (2.75)
  Post-Operative Day 1, after noon | 2.52 (1.88) | 3.65 (2.6)
  Post-Operative Day 2, midnight | 2.19 (1.86) | 3.83 (2.58)
  Post-Operative Day 2, before noon | 1.94 (1.42) | 3.77 (2.94)
  Post-Operative Day 2, after noon | 1.81 (1.43) | 3.5 (2.52)
  Post-Operative Day 3, before noon | 1.57 (1.55) | 3.16 (2.39)
  Post-Operative Day 3, after noon | 1.56 (1.51) | 2.98 (2.39)
  Post-Operative Day 4, before noon | 1.14 (1.19) | 2.44 (2.02)
  Post-Operative Day 4, after noon | 1.29 (1.47) | 2.93 (2.58)
  Post-Operative Day 5, before noon | 1.64 (1.88) | 2.54 (1.88)
  Post-Operative Day 5, after noon | 1.48 (1.8) | 2.79 (2.14)
  Post-Operative Day 6, before noon | 1.56 (2.41) | 2.26 (2.11)
  Post-Operative Day 6, after noon | 1.41 (2.34) | 2.50 (2.19)
  Post-Operative Day 7, before noon | 1.36 (2.38) | 2.25 (2.14)
  Post-Operative Day 7, after noon | .99 (1.4) | 2.12 (2.24)
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; Mean NRS-11 score at post-operative day 7 (compared between the two arms); Test type: Superiority; p = 0.01, t-test, 2 sided; Mean Difference (Final Values) = -1.13, 95% CI 2-sided [-2.02 to -0.24] — Direction of mean difference is Gabapentin arm minus placebo arm

2. Secondary Outcome: Opioid Consumption, as Measured by Number of Tablets Taken.
Description: Participants were requested to self-report the number of opioid tablets (oxycodone, 5mg) that they had taken since the last survey.
Time Frame: Post-operative day 0 (the day of surgery, after surgery was completed) through post-operative day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of oxycodone 5mg tablets consumed
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 35 | 35
Number of oxycodone 5mg tablets consumed
  Post-Operative Day 0 | 1.11 (.32) | 1.54 (1.31)
  Post-Operative Day 1, midnight | 1.14 (.43) | 1.24 (.74)
  Post-Operative Day 1, before noon | 1.2 (.47) | 1.38 (.98)
  Post-Operative Day 1, after noon | 1.14 (.36) | 1.27 (.52)
  Post-Operative Day 2, midnight | 1.18 (.39) | 1.23 (.63)
  Post-Operative Day 2, before noon | 1.18 (.52) | 1.48 (1.06)
  Post-Operative Day 2, after noon | 1.12 (.33) | 1.52 (1.7)
  Post-Operative Day 3, before noon | 1.09 (.29) | 1.2 (.48)
  Post-Operative Day 3, after noon | 1.09 (0.29) | 1.11 (0.32)
  Post-Operative Day 4, before noon | 1.06 (0.24) | 1.10 (0.31)
  Post-Operative Day 4, after noon | 1.03 (0.17) | 1.00 (0.00)
  Post-Operative Day 5, before noon | 1.00 (0.00) | 1.00 (0.00)
  Post-Operative Day 5, after noon | 1.07 (0.26) | 1.08 (0.28)
  Post-Operative Day 6, before noon | 1.00 (0.00) | 1.12 (0.33)
  Post-Operative Day 6, after noon | 1.00 (0.00) | 1.04 (0.20)
  Post-Operative Day 7, before noon | 1 (0) | 1.05 (.21)
  Post-Operative Day 7, after noon | 1 (0) | 1.05 (.22)
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; Mean number of opioid tablets taken at post-operative day 7 (compared between the two arms); Test type: Superiority; p = 0.19, t-test, 2 sided; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.13 to 0.03] — Direction of mean difference is Gabapentin arm minus placebo arm

3. Secondary Outcome: Change in Narcotic Consumption, as Measured by Frequency of Narcotic Tablets Taken
Description: Frequency of narcotic tablets that were taken after surgery
Time Frame: Post-operative day 0 (the day of surgery, after surgery was completed) through post-operative day 7
Population: Data was not collected for this measure.
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Narcotic Consumption, as Measured by Duration of Narcotic Tablets Consumption
Description: Duration (time period) over which narcotic tablets that were consumed
Time Frame: Post-operative day 0 (the day of surgery, after surgery was completed) through post-operative day 7
Population: Data was not collected for this measure.
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: After surgery (post-operative day 0) through 2 weeks post-operatively.
Description: Adverse events were self-reported by participants from the day of surgery (post-operative day 0) through post-operative day 7, along with pain score and number of opioid tablets taken. Participants were also evaluated and assessed for adverse events 2-weeks post-operatively by the surgeon.
Arm/Group | Gabapentin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/36 | 2/38
Other Adverse Events (participants affected / at risk) | 16/36 | 15/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin (N=36) | Placebo (N=38)
syncopal episode (General disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin (N=36) | Placebo (N=38)
GI upset (abdominal pain, bloating, heartburn) (Gastrointestinal disorders) | 4 (4) | 9 (9)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Paresthesia (Nervous system disorders) | 5 (5) | 3 (3)
Blurry vision (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Dizziness (General disorders) | 5 (5) | 1 (1)
Lightheadedness (General disorders) | 1 (1) | 3 (3)
Somnolence, drowsiness (General disorders) | 4 (4) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Insomnia (General disorders) | 1 (1) | 1 (1)
Hot flashes (General disorders) | 0 (0) | 1 (1)
Weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT04230980/Prot_SAP_000.pdf